CLINICAL TRIAL: NCT05908877
Title: Complex Assessment and Monitoring of Cardio-metabolic Risk in Overweight and Obese Children
Brief Title: Cardio-Metabolic Risk Evaluation in Overweight and Obese Children
Acronym: CardMetSOb
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Neoped - Centru de Pediatrie (Other)
Collaborators: University of Medicine and Pharmacy "Victor Babes" Timisoara (Other); West University of Timisoara (Other)
Responsible Party: Principal Investigator, Teofana-Otilia Bizerea-Moga, Teaching Assistant, University of Medicine and Pharmacy "Victor Babes" Timisoara
Other Study IDs: 01:Cardio_MetS_Ob
Record Dates: First submitted 2022-12-04; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Pediatric Obesity; Metabolic Syndrome; Nonalcoholic Fatty Liver; Atherosclerosis; Psychology; Cardiometabolic Syndrome
Keywords: Pediatric MetS, NAFLD, CIMT, Nutrition, Psychology
MeSH Terms: conditions — Pediatric Obesity; Metabolic Syndrome; Non-alcoholic Fatty Liver Disease; Atherosclerosis | interventions — Health Records, Personal; Nutrition Assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Overweight and Obese Children: Children diagnosed as overweight or obese, defined by the Centers for Disease Control and Prevention (CDC) as a BMI between the 85th and 95th percentile, or above the 95th percentile for the same age and sex, respectively.
  Interventions: Other: History and Clinical evaluation; Diagnostic Test: Biological evaluation of the metabolic syndrome and components; Diagnostic Test: Ultrasound evaluation of subclinical atherosclerosis and visceral fat storage; Other: Nutritional assessment; Behavioral: Psychological evaluation of the impact of obesity/overweight

INTERVENTIONS:
Other: History and Clinical evaluation — HISTORY and CLINICAL EVALUATION and recording of the following parameters:
  * Gestational Age
  * Birth Weight
  * Gender
  * Weaning habits
  * Anthropometric indices: actual age; actual weight; actual height; body mass index BMI (kg/m2) + percentile; waist circumference; age for height; weight for height; height for age; height standard deviation score (SDS)
  * Vital parameters: heart rate (beats/min); respiratory rate (breaths/min); blood pressure (mmHg)
  * Adipose tissue
  * Subcutaneous fat tissue distribution
  * Acanthosis Nigricans
  * Stretch marks (striae)
  * Tanner Puberty Stage
Diagnostic Test: Biological evaluation of the metabolic syndrome and components — LABORATORY INVESTIGATIONS will include:
  * Lipid Profile: total cholesterol (mmol/L); LDL - cholesterol (mmol/L); HDL - cholesterol (mmol/L); triglycerides (mmol/L)
  * Glucose - Insulin Profile: HbA1c (%); serum glucose (mmol/L); insulinemia (µUI/mL); HOMA Index
  * Liver Function: alanine aminotransferase (ALT or TGP) (U/L); gamma glutamyl transferase (GGT) (U/L)
  * Cardio-Vascular Risk - Inflammation - Oxidative Stress: ultrasensitive C-reactive protein (ng/mL); leptin (ng/mL); adiponectin (ng/mL); serum selenium (μg/L); glutathione peroxidase (GPx) (U/L)
Diagnostic Test: Ultrasound evaluation of subclinical atherosclerosis and visceral fat storage — ULTRASOUND EVALUATION by:
  * Carotid Intima-Media Thickness (cIMT) Measurement using B-Mode ultrasound (Samsung Medison UGEO H60 Ultrasound System, Samsung Medison CO., LTD., Seoul Korea) with a high frequency linear array probe (5-13 MHz) and a semi-automated software (Auto IMT+), according to the Mannheim Consensus
  * Measurements of Visceral-to-Subcutaneous-Fat Ratio using B-Mode ultrasound (Samsung Medison UGEO H60 Ultrasound System, Samsung Medison CO., LTD., Seoul Korea) with a 7.5 (12) MHz linear transducer for subcutaneous fat and a 3.5 MHz convex transducer for visceral fat measurement
  * Ultrasound Quantification of Hepatic Steatosis: assessed with B-Mode ultrasound (Samsung Medison UGEO H60 Ultrasound System, Samsung Medison CO., LTD., Seoul Korea) using 3.5 MHz convex transducer; increased liver echogenicity, blurring of vascular margins and increased acoustic attenuation are the parameters considered in the quantification of hepatic steatosis
Other: Nutritional assessment — NUTRITION CONSULT Initial consult will include: food habits survey aiming at identifying the nutritional factors that led to an increased Body Mass Index (BMI) and recommendations At reevaluations the food diary of the patients will be evaluated and recommendations will be adapted accordingly.
  The final visit will include evaluation of the food diary looking to identify the factors that have or have not helped to normalize BMI in order to recommend a long-term healthy lifestyle.
Behavioral: Psychological evaluation of the impact of obesity/overweight — PSYCHOLOGICAL ASSESSMENT by:
  Evaluation of pediatric health-related quality of life will be assessed with Pediatric Quality of Life Inventory (PedsQL). The questionnaire has 23 items and undertakes the four types of functioning: physical, emotional, social, and educational. It can be filled in by children as well as parents. Higher scores indicate better health-related quality of life.
  Another questionnaire that will be used is the the Rosenberg Self-Esteem Scale. It is composed of 10 questions and measures positive and negative feelings about the self. The answer range is from strongly agree to strongly disagree. A higher score means higher self-esteem.
  Drawing in children is a communicative tool, many times more than reading or language. It can measure the image of the self and the image of the others and is representative of the unconscious.
  Questionnaires and drawing interpretation will be done at the initial presentation and at every control visit.

SUMMARY:
Metabolic and cardio-vascular complications can often appear in overweight and obese children from an early age. Currently, there are few studies in the specialized literature that correlate clinical, biological and ultrasound parameters in order to stratify cardio-metabolic risk in obese children. Also, the specialized literature is poor regarding longitudinal follow-up and the importance of diet for reducing metabolic and cardiovascular complications in these children.

This study is designed to assess the hypothesis that the sustained improvement of lifestyle with regard to nutrition and exercise can reverse cardiometabolic multimorbidities in obese children as assessed by clinical, biological and ultrasound evaluation.

DETAILED DESCRIPTION:
The Metabolic Syndrome (MetS) is a group of metabolic conditions that increase the risk of cardiovascular events, insulin resistance and type 2 diabetes. Obesity is often the first stage in the subsequent development of MetS. Further, one or more changes may occur, such as: an increase in triglycerides, low-density lipoprotein cholesterol (LDL-C), insulin resistance and blood pressure, respectively a decrease in high-density lipoprotein cholesterol (HDL-C) and glucose tolerance.

The term "nonalcoholic fatty liver disease" (NAFLD) refers to a spectrum of conditions ranging from steatosis to nonalcoholic steatohepatitis (NASH) and fibrosis rather than a single entity. The main risk factors are obesity and the metabolic dysregulations that it causes. Obesity contributes to the development of NAFLD because it not only leads to metabolic imbalance but also increases oxidative stress and mitochondrial dysfunction.

An early indication of metabolic and cardiovascular subclinical disease, is represented by an increase of the carotid intima-media thickness (CIMT), of subcutaneous and visceral adipose tissue, as well as the fatty liver deposition. B-mode ultrasound allows measuring of all these parameters thereby contributing to the early detection of changes at these levels.

The ever-increasing incidence of pediatric obesity, enhanced by the recent coronavirus (COVID-19) pandemic, imposes the need for clinical, paraclinical-imaging, biological, nutritional and psychological evaluation and monitoring of this population.

The study aims to develop an algorithm for the complex assessment of cardio-metabolic risk in overweight and obese children on the one hand, as well as to reduce this risk by establishing a nutrition and physical activity plan simultaneously with a continuous monitoring of the results obtained following this plan, on the other side.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of overweight or obesity
* informed consent of caregivers

Exclusion Criteria:

* lean/normal weight subjects
* monogenic or syndromic obesity
* endocrine obesity (e.g., hypothyroidism, Cushing's syndrome)
* medication-induced obesity
* associated chronic diseases (other than components of the metabolic syndrome)
* lack of informed consent of caregivers

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The group or cohort of patients will be selected form the population that addresses the primary care clinic - pediatric center - Neoped.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-07-10 (Estimated); Primary Completion 2023-12-10 (Estimated); Study Completion 2024-07-10 (Estimated)

PRIMARY OUTCOMES:
Changes from Baseline Body Mass Index in Overweight or Obese Children after Physical Activity and Diet Interventions | 0,3,6 and 12 months
  Initial measurement of the body mass index (BMI) followed by three additional measurements at 3,6 and 12 months will be performed. These aim to assess the changes from baseline body mass index (BMI) in overweight or obese children, after physical activity and diet interventions.
  Overweight and obesity are defined using age-specific BMI reference guidelines from the 2000 Centers for Disease Control and Prevention Child Growth Charts. Thus, overweight assumes BMI values between the 85th and 95th percentiles, and obesity implies values above the 95th percentile.
Changes from Baseline Systolic Blood Pressure in Overweight or Obese Children after Physical Activity and Diet Interventions | 0,3,6 and 12 months
  Initial evaluation of systolic blood pressure followed by three reevaluations at 3,6 and 12 months will be performed. These aim to assess the changes from baseline systolic blood pressure in overweight or obese children, after physical activity and diet interventions.
  Arterial hypertension is diagnosed as a blood pressure value (systolic, diastolic or both), measured in mmHg, over the 95th percentile for age.
Changes from Baseline Diastolic Blood Pressure in Overweight or Obese Children after Physical Activity and Diet Interventions | 0,3,6 and 12 months
  Initial evaluation of diastolic blood pressure followed by three reevaluations at 3,6 and 12 months will be performed. These aim to assess the changes from baseline diastolic blood pressure in overweight or obese children after physical activity and diet interventions.
  Arterial hypertension is diagnosed as a blood pressure value (systolic, diastolic or both), measured in mmHg, over the 95th percentile for age.
Evaluation of Changes in Health-Related Quality of Life in Children diagnosed with Overweight or Obesity after Physical Activity and Diet Interventions, using the Pediatric Quality of Life Inventory (PedsQL) | 0,6 and 12 months
  The questionnaire has 23 items and undertakes the four types of functioning: physical, emotional, social, and educational. It can be filled in by children as well as parents. Higher scores indicate better health-related quality of life.
  PedsQL will be used at the child's first assessment and reapplied at each control visit.
  Items on the PedsQL Generic Core Scales are reverse scored and transformed to a 0-100 scale. Higher scores indicate better health related quality of life:
  0 ("Never") = 100
  1. ("Almost Never") = 75
  2. ("Sometimes") = 50
  3. ("Often") = 25
  4. ("Almost Always") = 0 Scale scores are computed as the sum of the items over the number of items answered (to account for missing data). If more than 50% of items or more are missing, the Scale Score should not be computed.
Evaluation of Changes in Individual Self-Esteem in Children diagnosed with Overweight or Obesity after Physical Activity and Diet Interventions, using the Rosenberg self-esteem scale | 0,6 and 12 months
  This scale is composed of 10 questions and measures positive and negative feelings about the self. The answer range is from strongly agree to strongly disagree.
  The scale ranges from 0-30. Scores between 15 and 25 are within normal range; scores below 15 suggest low self-esteem.

SECONDARY OUTCOMES:
Ultrasound Evaluation of Changes in Liver Echogenicity in Children diagnosed with Overweight or Obesity after Physical Activity and Diet Interventions | 0,3,6 and 12 months
  Initial ultrasound evaluation of liver echogenicity followed by three reevaluations at 3,6 and 12 months will be performed. These aim to assess changes in liver echogenicity and the reduction in hepatic steatosis grade, if diagnosed at onset, in overweight or obese children after physical activity and diet interventions.
  Non-Alcoholic Fatty Liver Disease (NAFLD) can be diagnosed on ultrasound based on some suggestive parameters: diffuse hyperechoic structure ("bright liver"), deep beam attenuation, liver-to-kidney contrast, bright vessel walls.
  Non-Alcoholic Fatty Liver Disease (NAFLD) classification:
  * Grade 1 (mild): diffuse increase in liver echogenicity, with normal visualization of intrahepatic vessels and of the diaphragm.
  * Grade 2 (moderate): blurred visualization of intrahepatic vessels and of the diaphragm.
  * Grade 3 (severe): intrahepatic vessels, diaphragm and the posterior region of the liver cannot be visualized.
Ultrasound Evaluation of Changes in Visceral-to-Subcutaneous-Fat Ratio in Children diagnosed with Overweight or Obesity after Physical Activity and Diet Interventions | 0,3,6 and 12 months
  Initial ultrasound measurement of visceral and subcutaneous fat followed by three reevaluations at 3,6 and 12 months will be performed. These aim to assess changes in visceral-to-subcutaneous-fat ratio in overweight or obese children after physical activity and diet interventions.
  Subcutaneous fat thickness (ScFT) is defined as the measurement from the skin-fat interface to the anterior aspect of the linea alba.
  Visceral fat thickness (VFT) is defined as the thickness from the linea alba to the anterior wall of the aorta.
Changes of Carotid Intima-Media Thickness (CIMT) in Children diagnosed with Overweight or Obesity after Physical Activity and Diet Interventions | 0,3,6 and 12 months
  Initial ultrasound measurement of the carotid intima-media thickness (CIMT) followed by three reevaluations at 3,6 and 12 months will be performed. These aim to assess changes in carotid intima-media thickness in overweight or obese children after physical activity and diet interventions.
  At every visit four measurements of CIMT at far wall of the common carotid artery, approximately 1 cm proximal to the bulb, in the end-diastolic phase (2 for the left and 2 for the right CCA) will be obtained.
Changes from Baseline Serum Glucose Levels in Overweight or Obese Children after Physical Activity and Diet Interventions | 0,3,6 and 12 months
  Initial evaluation of glucose levels followed by three reevaluations at 3,6 and 12 months will be performed. These aim to assess the changes from baseline serum glucose levels in overweight or obese children after physical activity and diet interventions.
  Impaired glucose metabolism is defined as serum insulin levels over 15 mU/L or fasting blood glucose levels higher than 6.11 mmol/L.
Changes from Baseline Serum Lipid Levels in Overweight or Obese Children after Physical Activity and Diet Interventions | 0,3,6 and 12 months
  Initial evaluation of serum lipid levels followed by three reevaluations at 3,6 and 12 months will be performed. These aim to assess the changes from baseline serum lipid levels in overweight or obese children after physical activity and diet interventions.
  Dyslipidemia is defined if triglyceride or total cholesterol levels exceed the 95th percentile for age and sex or if or high-density lipoprotein (HDL) cholesterol levels are below the 5th percentile for age and sex.
Changes from Baseline Liver Function Tests in Overweight or Obese Children after Physical Activity and Diet Interventions | 0,3,6 and 12 months
  Liver function will be assessed by determining serum levels of alanine aminotransferase (ALT or TGP) (U/L) and gamma glutamyl transferase (GGT) (U/L) at the initial evaluation, and again at 3, 6 and 12 months. The aim is to assess the changes from baseline ALT and GGT levels in overweight or obese children after physical activity and diet interventions.
Changes from Baseline Serum Insulin Levels in Overweight or Obese Children after Physical Activity and Diet Interventions | 0,3,6 and 12 months
  Initial evaluation of serum insulin levels followed by three reevaluations at 3,6 and 12 months will be performed. These aim to assess the changes from baseline serum insulin levels in overweight or obese children after physical activity and diet interventions.
  In this study, IR will be evaluated by using the homeostasis model assessment for IR index (HOMA - IR), calculated using the following equation: HOMA - IR = fasting insulin (uU/mL) x fasting plasma glucose (mmol/L)/22.5.
  IR is diagnosed in a patient if HOMA-IR exceeds the 95th percentile for age and sex.
Changes from Baseline Inflammatory and Oxidative Stress Markers in Overweight or Obese Children after Physical Activity and Diet Interventions | 0,3,6 and 12 months
  Initial evaluation of inflammation and oxidative stress status by determining the serum levels of ultrasensitive C-reactive protein (ng/mL), leptin (ng/mL), adiponectin (ng/mL), selenium (μg/L) and glutathione peroxidase (GPx) (U/L). These parameters will be reevaluated at 3,6 and 12 months to assess the changes from baseline levels in overweight or obese children after physical activity and diet interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Teofana O Bizerea-Moga, MD PhD, Principal Investigator — Neoped - Centru de Pediatrie; "Victor Babeș" University of Medicine and Pharmacy Timișoara, Romania
Locations (1):
- Neoped - Centru de Pediatrie, Timișoara, Timiș County, Romania

IPD SHARING:
Plan to Share IPD: Undecided